CLINICAL TRIAL: NCT00692211
Title: Interventions to Improve Colorectal Cancer Screening Rates and Adherence
Brief Title: Interventions to Improve Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: SHP 08-177
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-04

CONDITIONS: Colorectal Neoplasms
Keywords: screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Fecal Immunochemical Tests (Experimental): Mailed fecal immunochemical tests
  Interventions: Other: Mailed fecal immunochemical tests
- Arm 2: Fecal Occult Blood Tests (Experimental): Mailed fecal occult blood tests
  Interventions: Other: Mailed fecal occult blood tests

INTERVENTIONS:
Other: Mailed fecal occult blood tests — Stool blood test
  Arms: Arm 2: Fecal Occult Blood Tests
Other: Mailed fecal immunochemical tests — Stool blood test
  Arms: Arm 1: Fecal Immunochemical Tests

SUMMARY:
We will evaluate if we can increase colorectal cancer screening rates by directly sending screening tests to patients rather than waiting for them to come to clinic visits. We are also evaluating a new test--fecal immunochemical tests--which does not require patients to make dietary or medication changes. We will see if patients are more likely to complete these tests than the standard fecal occult blood tests.

DETAILED DESCRIPTION:
Background: Colorectal cancer causes a substantial burden of suffering in the elderly VA population. Although colorectal cancer screening can reduce both the incidence and mortality from colorectal cancer, screening rates are low for the New Mexico VA Health Care System.

Objectives: We propose to use the electronic medical record and a new technology for fecal stool testing to improve screening rates and adherence to screening.

Methods: The electronic medical record will be used to identify patients who are eligible for screening but who do not have an immediately upcoming primary care clinic appointment. We will enroll a randomly-selected sample of 800 of these patients who have agreed to participate in the study and mail them stool tests along with instructions and educational information about the benefits of screening. We will compare the proportion of subjects who undergo colorectal cancer screening during the 3-month study period against a randomly-selected sample of 400 eligible patients who will require a clinic visit to initiate screening. Because adherence for fecal occult blood tests is low, we also propose to evaluate a new screening technology--fecal immunochemical stool tests which target intact human hemoglobin. These tests can be performed without requiring patients to follow onerous dietary and medication restrictions. We will evaluate whether screening adherence (proportion completing testing) is higher with fecal immunochemical testing (n = 400) compared to the standard fecal occult blood test (n=400). We will also evaluate the yield of advanced neoplasia for each of the screening tests.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for stool-based colorectal cancer screening, followed in primary care clinic

Exclusion Criteria:

* Need for surveillance or screening colonoscopy
* limited life expectancy

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2008-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Hoffman, MD, Principal Investigator — New Mexico VA Health Care System, Albuquerque, NM
Locations (1):
- New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico, United States

REFERENCES:
- [Result] Hoffman RM, Steel SR, Yee EF, Massie L, Schrader RM, Moffett ML, Murata GH. A system-based intervention to improve colorectal cancer screening uptake. Am J Manag Care. 2011 Jan;17(1):49-55. PMID 21348568
- [Result] Hoffman RM, Steel S, Yee EF, Massie L, Schrader RM, Murata GH. Colorectal cancer screening adherence is higher with fecal immunochemical tests than guaiac-based fecal occult blood tests: a randomized, controlled trial. Prev Med. 2010 May-Jun;50(5-6):297-9. doi: 10.1016/j.ypmed.2010.03.010. Epub 2010 Mar 20. PMID 20307568

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Fecal Immunochemical Tests: Mailed fecal immunochemical tests
  Fecal immunochemical testing: Stool blood test
- Arm 2: Fecal Occult Blood Tests: Mailed fecal occult blood tests
  Fecal occult blood test: Stool blood test
Period: Overall Study
Arm/Group | Arm 1: Fecal Immunochemical Tests | Arm 2: Fecal Occult Blood Tests
Started | 202 | 202
Completed | 202 | 202
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Fecal Immunochemical Tests | Arm 2: Fecal Occult Blood Tests | Total
Number analyzed (Participants) | 202 | 202 | 404
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 128 | 131 | 259
  >=65 years | 74 | 71 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (7.3) | 63.9 (8.1) | 63.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 12
  Male | 199 | 193 | 392
Region of Enrollment [Number; unit: participants]
  United States | 202 | 202 | 404

OUTCOME MEASURES:

1. Primary Outcome: Colorectal Cancer Screening
Description: Completing fecal blood test within 90 days of enrolling
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Arm 1: Fecal Immunochemical Tests | Arm 2: Fecal Occult Blood Tests
Number analyzed (Participants) | 202 | 202
participants | 127 | 112
Statistical Analysis 1: Comparison: Arm 1: Fecal Immunochemical Tests vs Arm 2: Fecal Occult Blood Tests; Study powered to detect 10% difference in proportion of screening adherence based on alpha of 0.05, beta 0.20; Test type: Superiority or Other; p = 0.01, Regression, Logistic — Not adjusted for multiple comparisons, a priori threshold of 0.05; Odds Ratio (OR) = 1.56, 95% CI 2-sided [1.04 to 2.32]

ADVERSE EVENTS:
Arm/Group | Arm 1: Fecal Immunochemical Tests | Arm 2: Fecal Occult Blood Tests
Serious Adverse Events (participants affected / at risk) | 0/202 | 0/202
Other Adverse Events (participants affected / at risk) | 0/202 | 0/202

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No